CLINICAL TRIAL: NCT03506737
Title: Impact of an Exercise-based Cardiac Rehabilitation Program on Hospitalized Heart Failure Patients Submitted to Cardiac Transplantation: Clinical Trial
Brief Title: Exercise-based Cardiac Rehabilitation Program on Hospitalized Heart Failure Patients Submitted to Cardiac Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Caroline Bublitz Barbosa, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 74619617.3.0000.5505
Record Dates: First submitted 2018-04-04; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure; Transplant; Failure, Heart; Physical Activity
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exercise protocol (Experimental): Conventional global exercise
  Interventions: Other: Conventional exercise protocol
- Cycle ergometer exercise protocol (Experimental): Stationary cycle ergometer exercise
  Interventions: Other: Cycle ergometer exercise protocol

INTERVENTIONS:
Other: Conventional exercise protocol — Breathing exercises and global active exercises of the upper and lower limbs while in the upright seated position
  Arms: Conventional exercise protocol
Other: Cycle ergometer exercise protocol — Stationary cycle ergometer exercise while in the upright seated position for 20 minutes. The protocol will be performed intermittently with 5 periods; each period consists of 3 minutes of cycling followed by 1-minute of rest.
  Arms: Cycle ergometer exercise protocol

SUMMARY:
Objective: To evaluate the effects of an early-based cardiac rehabilitation program on the functional capacity, inspiratory muscular strength and clinical outcomes in hospitalized heart failure patients before and after heart transplantation. Method: 30 hospitalized heart failure patients awaiting cardiac transplantation will be selected and randomized in 2 groups: conventional group (n = 15) - conventional exercise protocol: breathing exercises and global active exercises of upper and lower limbs in the sitting position; and Intervention group (n = 15) - cycle ergometer exercise protocol: each session consists of cycling on a stationary bicycle in the seated position for 20 minutes. In both groups, the exercise protocols will be applied twice a day until the hospital discharge, always supervised by a physiotherapist and a doctor. The evaluation procedures in all patients of the research will be: functional capacity measured by the 6 minute walk test and inspiratory muscle strength measured by manovacuometry. Evaluations will be repeated in 3 distinct moments: after 24h of hospital admission and/or clinical stabilization; before transplantation and after transplantation in hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure diagnosis determined by clinical presentation and confirmed on echocardiography by clinicians, with a left ventricular ejection fraction (LVEF) < 40%
* New York Heart Association (NYHA) classes III and IV.

Exclusion Criteria:

* chronic lung disease confirmed by pulmonary function testing
* unstable angina pectoris and acute coronary syndromes
* dialysis
* neuromuscular and psychiatric conditions that interfere in exercise

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test to measure functional capacity change | After 24 hours of hospital admission or clinical stabilization; before transplantation (after 4 weeks of rehabilitation program) and in hospital discharge (after 4 weeks of transplantation).
  According to the baseline distance walked, we will evaluate the improvement in functional capacity after the period of the rehabilitation programs
Respiratory muscle strength | After 24 hours of hospital admission or clinical stabilization; before transplantation (after 4 weeks of rehabilitation program) and in hospital discharge (after 4 weeks of transplantation)
  By manovacuometry, assessing the change in inspiratory muscle pressure and expiratory muscle pressure

SECONDARY OUTCOMES:
Invasive mechanical ventilation | First day after transplantation.
  Duration of invasive mechanical ventilation will be recorded after cardiac transplantation.
Duration of intensive care unit stay | In hospital discharge (after 4 weeks of transplantation).
  Duration of stay in intensive care unit (in days) after transplantation will be recorded.
Hospitalization stay | In hospital discharge (after 4 weeks of transplantation).
  Duration of stay in the hospital (in days) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Caroline Bublitz Barbosa, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No